CLINICAL TRIAL: NCT05758402
Title: A Randomized, Open, Parallel, Controlled, Multi-center, Interventional, Cross-sectional Study to Evaluate the Detection Rate of Psoriatic Arthritis in Korean Moderate-to-severe Psoriasis Patients, With or Without Active Screening for Arthritis in Psoriasis (ASAP Study)
Acronym: ASAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAIN457AKR04
Record Dates: First submitted 2023-01-09; First posted 2023-03-07 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: Psoriatic arthritis; PsA; Psoriasis; PsO; Early arthritis for psoriatic patients; EARP; Classification criteria for psoriatic arthritis; CASPAR
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EARP group (Other): For the EARP group, the investigator provided this questionnaire to participants, who filled out it based on their symptoms. Afterwards, the investigator calculated the total score of the questionnaire answered by the participant, and further evaluated the participants using the CASPAR.
  Interventions: Diagnostic Test: EARP group
- Routine practice group (Active Comparator): In the control group, PsA risk was assessed in moderate to severe PsO patients as per routine practice without using the EARP screening. After the completion of PsA risk assessment via routine practice according to the investigator's judgement, the participants were further evaluated using the CASPAR.
  Interventions: Diagnostic Test: Routine practice group

INTERVENTIONS:
Diagnostic Test: Routine practice group — Routine practice group
  Arms: Routine practice group
Diagnostic Test: EARP group — EARP group
  Arms: EARP group

SUMMARY:
This was a randomized, open, parallel, controlled, multi-center, interventional, cross-sectional study to evaluate the detection rate of Psoriatic arthritis (PsA) in Korean moderate to severe Psoriasis (PsO) patients with or without the Early arthritis for psoriatic patients (EARP) screening.

DETAILED DESCRIPTION:
All procedures for each patient were performed for one day. If an additional time was required depending on the circumstances of the institution and so on, the data specified in this study protocol were recommended to be collected as soon as possible. After the participants enrolled in this study, they were assessed whether they met the inclusion/exclusion criteria. In terms of the severity of PsO, it was assessed with the Psoriasis Area and Severity Index (PASI) and if the score of 10 or higher was defined as moderate to severe PsO. A total 368 eligible participants were randomized 1:1 ratio into the EARP group and the Routine practice group.

For the EARP group, the investigator asked the participants about the EARP questionnaire consisting of 10 questions. When the EARP score >= 3, the participants were suspected for having potential PsA. For Routine practice group, the investigator selected the participants suspected of PsA in consideration of the various clinical characteristics of the participants.

After the completion of EARP questionnaire evaluation and the investigator's judgement as per routine practice in each group, all the participants were evaluated using Classification criteria for psoriatic arthritis (CASPAR). According to the CASPAR, participants having inflammatory articular disease with 3 or more points from the CASPAR were diagnosed as PsA, and the detection rate of PsA in each group was evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is >= 19 years of age at the time of study enrollment
* Patient who had an established diagnosis of PsO based upon clinical evidence and documented medical history
* Patient who is moderate to severe PsO (Psoriasis Area and Severity Index (PASI) score >= 10)
* Patient who is willing and able to comply with study procedures
* Patient who is able to provide the informed consent form (ICF)

Exclusion Criteria:

* Patients who have formal pre-existing diagnosis of PsA
* Patients who have ever received treatment with biologic Disease-Modifying Anti-Rheumatic Drugs (DMARDs)
* Patients who currently receive systemic glucocorticoids
* Patients who currently receive opioid analgesics
* Patients who has other known pre-existing dermatological or rheumatological diseases:

  * Non-plaque psoriasis
  * Rheumatoid arthritis
  * Osteoarthritis
  * Gout
  * Reactive arthritis
  * Ankylosing spondylitis
  * Axial spondyloarthritis
  * Enteropathic arthritis
  * Plantar fasciitis
  * Systemic lupus erythematosus (SLE)
* Female patients who are pregnant
* Patients who are participating in other interventional clinical trials
* Patients who have already had PsA screening via screening questionnaires or imaging

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- South Korea (8):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Bucheon-si
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 15 centers in the Republic of Korea.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were centrally, randomly allocated with a 1:1 ratio to either the EARP group or the Routine practice group using an Interactive Web Response System (IWRS).
Period: Overall Study
Arm/Group | EARP Group | Routine Practice Group
Started (All enrolled participants were included in the Full Analysis Set (FAS)) | 181 | 187
Completed | 181 | 187
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EARP Group | Routine Practice Group | Total
Number analyzed (Participants) | 181 | 187 | 368
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.22 (15.00) | 43.48 (14.11) | 44.33 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 35 | 99
  Male | 117 | 152 | 269
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 181 | 187 | 368
Height [Mean (Standard Deviation); unit: cm] | 169.07 (8.87) | 171.48 (8.58) | 170.29 (8.80)
Weight [Mean (Standard Deviation); unit: kg] | 74.41 (16.54) | 75.53 (15.66) | 74.98 (16.09)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.87 (4.65) | 25.54 (4.38) | 25.70 (4.51)
Drinking history [Count of Participants; unit: Participants]
  Current | 99 | 107 | 206
  Past | 47 | 46 | 93
  Never | 35 | 34 | 69
Smoking history [Count of Participants; unit: Participants]
  Current | 80 | 91 | 171
  Past | 30 | 29 | 59
  Never | 71 | 67 | 138
Duration of Psoriasis (PsO) [Mean (Standard Deviation); unit: months] | 124.33 (129.16) | 114.20 (126.14) | 119.19 (127.56)
Psoriasis Area and Severity Index (PASI) score [Mean (Standard Deviation); unit: Unit on a scale] — PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). The body is divided into four sections (head (H) (10% of a person's skin); arms (A) (20%); trunk (T) (30%); legs (L) (40%)). Each of these areas is scored by itself, and then the four scores are combined into the final PASI.
  Unit on a scale | 13.55 (4.78) | 13.70 (4.98) | 13.63 (4.88)
Psoriasis Area and Severity Index (PASI) category [Count of Participants; unit: Participants] — PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). The body is divided into four sections (head (H) (10% of a person's skin); arms (A) (20%); trunk (T) (30%); legs (L) (40%)). Each of these areas is scored by itself, and then the four scores are combined into the final PASI.
  Participants
    10 to <12 | 93 | 98 | 191
    12 to <14 | 39 | 33 | 72
    14 to <16 | 13 | 21 | 34
    16 to <18 | 14 | 15 | 29
    18 to <20 | 5 | 2 | 7
    >= 20 | 17 | 18 | 35
Psoriasis (PsO) family history [Count of Participants; unit: Participants]
  Yes | 26 | 28 | 54
  No | 155 | 159 | 314
Psoriatic Arthritis (PsA) family history [Count of Participants; unit: Participants]
  Yes | 4 | 0 | 4
  No | 177 | 187 | 364
Presence or absence of hard-to-treat area involvement (scalp, palmoplantar, nails) [Count of Participants; unit: Participants]
  Yes | 117 | 121 | 238
  No | 64 | 66 | 130
Presence or absence of musculoskeletal symptoms [Count of Participants; unit: Participants]
  Yes | 42 | 44 | 86
  No | 139 | 143 | 282
Total Nail Psoriasis Severity Index (NAPSI) score [Mean (Standard Deviation); unit: Unit on a scale] — The Nail Psoriasis Severity Index (NAPSI) score is used to measure psoriasis of the nails. Each nail is divided into 4 equal and symmetrical quadrants to properly assess nail matrix and nail bed changes. Each nail is given a score for nail bed PsO and nail matrix PsO ranging from 0 (none) to 4 (present in 4/4 nail) depending on the presence of any of the features of nail PsO in that quadrant. A total score per nail is 0-8, and the range of the total scores from all nails is 0-160 (toenails are included).
  Unit on a scale
    NAPSI score of left hand | 4.71 (7.91) | 5.56 (9.14) | 5.14 (8.55)
    NAPSI score of right hand | 4.61 (7.94) | 5.85 (9.68) | 5.24 (8.88)
    NAPSI score of left foot | 3.71 (8.30) | 5.71 (10.35) | 4.73 (9.44)
    NAPSI score of right foot | 4.01 (8.10) | 5.95 (10.46) | 4.99 (9.41)
    Total NAPSI score | 17.04 (29.14) | 23.06 (36.70) | 20.10 (33.29)
SJC66/TJC68 total joint count [Mean (Standard Deviation); unit: Joint count] — 66 swollen and 68 tender joints are assessed (the hips are not assessed for swelling). The joint count is scored as a sum of the tender joints and a sum of the swollen joints. SJC66: swollen joint count in 66 joints; TJC68: tender joint count in 66 joints.
  Joint count
    SJC66 joint count | 1.00 (4.89) | 0.77 (4.45) | 0.88 (4.67)
    TJC68 joint count | 1.32 (4.53) | 1.12 (4.55) | 1.22 (4.54)
    SJC66/TJC68 total joint count | 2.32 (8.97) | 1.89 (8.53) | 2.10 (8.74)

OUTCOME MEASURES:

1. Primary Outcome: Detection Rate of Psoriatic Arthritis (PsA)
Description: After the completion of EARP questionnaire evaluation and the investigator's judgement as per routine practice in each group, all the participants were evaluated using Classification criteria for psoriatic arthritis (CASPAR). According to the CASPAR, participants having inflammatory articular disease with 3 or more points from the CASPAR were diagnosed as PsA, and the detection rate of PsA in each group was evaluated and compared.
  The detection rate of Psoriatic Arthritis (PsA) amongst moderate to severe Psoriasis (PsO) patients between the EARP group and the Routine practice groups was defined as the percentage of patients with true positive results divided by all patients in each EARP and Routine practice group.
  The true positive results were defined as patients with a classification criteria for psoriatic arthritis (CASPAR) score >= 3 among EARP >= 3 for the EARP group and among those suspected of PsA by investigator's judgement for the Routine Practice group.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | EARP Group | Routine Practice Group
Number analyzed (Participants) | 181 | 187
Participants | 8 | 6
Statistical Analysis 1: Comparison: EARP Group vs Routine Practice Group; Test type: Other; p = 0.544, Chi-squared; Rate difference = 1.21, 95% CI 2-sided [-2.71 to 5.13] — Rate difference = detection rate of PsA in EARP group - detection rate of PsA in routine practice group

2. Secondary Outcome: Sensitivity, Specificity, Positive Predictive Value (PPV) and Negative Predictive Value (NPV) Between EARP Questionnaire (EARP Group) and the Investigator's Judgement (Routine Practice Group)
Description: Sensitivity was summarized with the number and percentage of patients who have true positive (TP) among those who have true positive (TP) and false negative (FN).
  Specificity was summarized with the number and percentage of patients who have true negative (TN) among those who have true negative (TN) and false positive (FP).
  Positive predictive value (PPV) was summarized with the number and percentage of patients who have true positive (TP) among those who have true positive (TP) and false positive (FP).
  Negative predictive value (NPV) was summarized with the number and percentage of patients who have true negative (TN) among those who have true negative (TN) and false negative (FN).
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | EARP Group | Routine Practice Group
Number analyzed (Participants) | 181 | 187
Participants
  Sensitivity: number analyzed (Participants) | 13 | 15
  Sensitivity | 8 | 6
  Specificity: number analyzed (Participants) | 168 | 172
  Specificity | 129 | 157
  Positive Predictive Value (PPV): number analyzed (Participants) | 47 | 21
  Positive Predictive Value (PPV) | 8 | 6
  Negative Predictive Value (NPV): number analyzed (Participants) | 134 | 166
  Negative Predictive Value (NPV) | 129 | 157
Statistical Analysis 1: Comparison: EARP Group vs Routine Practice Group; Sensitivity; Test type: Other; p = 0.256, Chi-squared
Statistical Analysis 2: Comparison: EARP Group vs Routine Practice Group; Specificity; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: EARP Group vs Routine Practice Group; Positive Predictive Value (PPV); Test type: Other; p = 0.336, Fisher Exact
Statistical Analysis 4: Comparison: EARP Group vs Routine Practice Group; Negative Predictive Value (NPV); Test type: Other; p = 0.490, Chi-squared

3. Secondary Outcome: Age Characteristics by Participants With or Without PsA
Description: Age characteristics between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Years
Groups:
- With PsA: Participants with PsA
- Without PsA: Participants without PsA
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Years | 48.14 (12.13) | 44.02 (14.71)
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Age characteristics; Test type: Other; p = 0.101, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Gender Characteristics by Participants With or Without PsA
Description: Gender characteristics between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Participants
  Male | 20 | 249
  Female | 8 | 91
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Gender characteristics; Test type: Other; p = 0.836, Chi-squared

5. Secondary Outcome: Body Mass Index (BMI) Characteristics by Participants With or Without PsA
Description: Body Mass Index (BMI) characteristics between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 339
kg/m^2 | 25.02 (3.38) | 25.76 (4.59)
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Body Mass Index (BMI) characteristics; Test type: Other; p = 0.520, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Drinking and Smoking History Characteristics by Participants With or Without PsA
Description: Drinking and smoking history characteristics between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Participants
  Drinking history: Current | 20 | 186
  Drinking history: Past | 4 | 89
  Drinking history: Never | 4 | 65
  Smoking history: Current | 12 | 159
  Smoking history: Past | 6 | 53
  Smoking history: Never | 10 | 128
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Drinking history characteristics; Test type: Other; p = 0.216, Chi-squared
Statistical Analysis 2: Comparison: With PsA vs Without PsA; Smoking history characteristics; Test type: Other; p = 0.719, Chi-squared

7. Secondary Outcome: Duration of Psoriasis (PsO) Characteristics by Participants With or Without PsA
Description: Duration of Psoriasis (PsO) characteristics between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: months
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
months | 132.08 (147.33) | 118.12 (125.99)
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Duration of Psoriasis (PsO) characteristics; Test type: Other; p = 0.831, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Family History of Psoriasis (PsO) and Psoriatic Arthritis (PsA) Characteristics by Participants With or Without PsA
Description: Family history of psoriasis (PsO) and psoriatic arthritis (PsA) characteristics between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Participants
  Psoriasis (PsO) family history: Yes | 6 | 48
  Psoriasis (PsO) family history: No | 22 | 292
  Psoriatic Arthritis (PsA) family history: Yes | 1 | 3
  Psoriatic Arthritis (PsA) family history: No | 27 | 337
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Family history of psoriasis (PsO) characteristics; Test type: Other; p = 0.274, Fisher Exact
Statistical Analysis 2: Comparison: With PsA vs Without PsA; Family history of psoriatic arthritis (PsA) characteristics; Test type: Other; p = 0.272, Fisher Exact

9. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score Characteristics by Participants With or Without PsA
Description: PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). The body is divided into four sections (head (H) (10% of a person's skin); arms (A) (20%); trunk (T) (30%); legs (L) (40%)). Each of these areas is scored by itself, and then the four scores are combined into the final PASI. For each section, the percent of area of skin involved, is estimated and then transformed into a grade from 0 (0% of involved area) to 6 (90-100% of involved area). Within each area, the severity is estimated by three clinical signs: erythema (redness), induration (thickness) and desquamation (scaling). Severity parameters are measured on a scale of 0 (none) to 4 (maximum). The sum of all three severity parameters is then calculated for each section of skin, multiplied by the area score for that area and multiplied by weight of respective section (0.1 for head, 0.2 for arms, 0.3 for body and 0.4 for legs).
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Unit on a scale | 13.76 (4.68) | 13.62 (4.90)
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Psoriasis Area and Severity Index (PASI) score characteristics; Test type: Other; p = 0.622, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: The Status of Hard-to-treat Area Involvement and Musculoskeletal Symptoms Characteristics by Participants With or Without PsA
Description: The presence or absence of hard-to-treat area involvement (scalp, palmoplantar, nails) and presence or absence of musculoskeletal symptoms between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Participants
  Presence or absence of hard-to-treat area involvement (scalp, palmoplantar, nails): Yes | 27 | 211
  Presence or absence of hard-to-treat area involvement (scalp, palmoplantar, nails): No | 1 | 129
  Presence or absence of musculoskeletal symptoms: Yes | 16 | 70
  Presence or absence of musculoskeletal symptoms: No | 12 | 270
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Status of hard-to-treat area involvement characteristics; Test type: Other; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: With PsA vs Without PsA; Status of musculoskeletal symptoms characteristics; Test type: Other; p < 0.001, Chi-squared

11. Secondary Outcome: Nail Psoriasis Severity Index (NAPSI) Score Characteristics by Participants With or Without PsA
Description: The Nail Psoriasis Severity Index (NAPSI) score is used to measure psoriasis of the nails. Each nail is divided into 4 equal and symmetrical quadrants to properly assess nail matrix and nail bed changes. Each nail is given a score for nail bed PsO and nail matrix PsO ranging from 0 (none) to 4 (present in 4/4 nail) depending on the presence of any of the features of nail PsO in that quadrant. A total score per nail is 0-8, and the range of the total scores from all nails is 0-160 (toenails are included).
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Unit on a scale
  NAPSI score of left hand | 10.43 (11.21) | 4.71 (8.17)
  NAPSI score of right hand | 9.18 (11.10) | 4.91 (8.61)
  NAPSI score of left foot | 9.29 (13.06) | 4.35 (9.00)
  NAPSI score of right foot | 9.54 (11.57) | 4.62 (9.13)
  Total NAPSI score | 38.43 (43.45) | 18.59 (31.93)
Statistical Analysis 1: Comparison: With PsA vs Without PsA; NAPSI score of left hand characteristics; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: With PsA vs Without PsA; NAPSI score of right hand characteristics; Test type: Other; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: With PsA vs Without PsA; NAPSI score of left foot characteristics; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: With PsA vs Without PsA; NAPSI score of right foot characteristics; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: With PsA vs Without PsA; Total NAPSI score characteristics; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: SJC66/TJC68 Total Joint Count Characteristics by Participants With or Without PsA
Description: 66 swollen and 68 tender joints are assessed (the hips are not assessed for swelling). The joint count is scored as a sum of the tender joints and a sum of the swollen joints. SJC66: swollen joint count in 66 joints; TJC68: tender joint count in 66 joints.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 54
Joint count
  SJC66 joint count | 5.36 (11.18) | 0.51 (3.44)
  TJC68 joint count | 6.00 (9.88) | 0.83 (3.53)
  SJC66/TJC68 total joint count | 11.36 (20.01) | 1.34 (6.57)
Statistical Analysis 1: Comparison: With PsA vs Without PsA; SJC66 total joint count characteristics; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: With PsA vs Without PsA; TJC68 total joint count characteristics; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: With PsA vs Without PsA; SJC66/TJC68 total joint count characteristics; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Solicited Medical History by Participants With or Without PsA
Description: The presence or absence of co-morbidities (heart diseases, stroke, diabetes, hyperlipidemia, hypertension and fatty liver)) between patients with PsA and without PsA were analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 28 | 340
Participants
  Heart diseases: Past | 0 | 0
  Heart diseases: Current | 3 | 8
  Heart diseases: Never | 25 | 332
  Stroke: Past | 0 | 0
  Stroke: Current | 0 | 3
  Stroke: Never | 28 | 337
  Diabetes: Past | 0 | 0
  Diabetes: Current | 2 | 27
  Diabetes: Never | 26 | 313
  Hyperlipidemia: Past | 0 | 0
  Hyperlipidemia: Current | 8 | 40
  Hyperlipidemia: Never | 20 | 300
  Hypertension: Past | 0 | 0
  Hypertension: Current | 9 | 62
  Hypertension: Never | 19 | 278
  Fatty liver: Past | 0 | 0
  Fatty liver: Current | 2 | 15
  Fatty liver: Never | 26 | 325
Statistical Analysis 1: Comparison: With PsA vs Without PsA; Heart diseases; Test type: Other; p = 0.043, Fisher Exact
Statistical Analysis 2: Comparison: With PsA vs Without PsA; Stroke; Test type: Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: With PsA vs Without PsA; Diabetes; Test type: Other; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: With PsA vs Without PsA; Hyperlipidemia; Test type: Other; p = 0.019, Chi-squared
Statistical Analysis 5: Comparison: With PsA vs Without PsA; Hypertension; Test type: Other; p = 0.073, Chi-squared
Statistical Analysis 6: Comparison: With PsA vs Without PsA; Fatty liver; Test type: Other; p = 0.377, Fisher Exact

14. Secondary Outcome: Percentage of Participants With PsO Related Treatment Other Than Medications by Participants With or Without PsA
Description: The presence or absence of PsO related treatment other than medications (UV light therapy, Psoralen with ultraviolet A (PUVA), Phototherapy and Laser therapy and Naturopathy) between patients with PsA and without PsA was analyzed and compared.
Time Frame: Visit 1 (Day 1)
Population: Full Analysis Set (FAS). Only participants with PsO related treatment other than medications included.
Measure: Count of Participants; unit: Participants
Arm/Group | With PsA | Without PsA
Number analyzed (Participants) | 3 | 40
Participants
  UV light therapy | 2 | 20
  Psoralen with ultraviolet A (PUVA) | 1 | 11
  Phototherapy | 0 | 7
  Laser therapy | 0 | 2

ADVERSE EVENTS:
Description: Safety evaluation was not applicable as no drug was involved.
Arm/Group | EARP Group | Routine Practice Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT05758402/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT05758402/SAP_001.pdf